CLINICAL TRIAL: NCT01854944
Title: PET Trial to Assess the Receptor Occupancy of Brexpiprazole in Adult Subjects With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331-09-219
Record Dates: First submitted 2013-05-07; First posted 2013-05-16 (Estimated); Results first posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brexpiprazole 1mg to 4mg (Experimental): Three cohorts of subjects will be evaluated:
  - Cohorts 1 and 3 will receive high doses of brexpiprazole, and Cohort 2 will receive low doses of brexpiprazole.
  Interventions: Drug: Brexpiprazole 1mg to 4mg

INTERVENTIONS:
Drug: Brexpiprazole 1mg to 4mg
  Other Names: Brexpiprazole

SUMMARY:
The purpose of this study is to determine how low and high does of brexpiprazole binds to certain receptors in the brain. This will be determined by PET scans taken pre-dose and post-dose.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Schizophrenia.
* Ability to provide written informed consent.
* Ability to understand the protocol and meet the protocol requirements.
* Must be in good physical health determined by ECG and laboratory values, medical history and physical examinations.
* Has stable disease, defined as meeting all of the following criteria: A CGI-S score <= 4 (moderately ill); A PANSS total score <= 60; A score of <= 4 (moderate) on any of the following PANSS items: (P7 (hostility); G8 (uncooperativeness)).
* Body mass index of 19 to 35 kg/m2

Exclusion Criteria:

* Sexually active males and females of childbearing potential who are not practicing double-barrier birth control, or who will not remain abstinent, during the trial and for 30 days following the last dose of trial medication. If employing birth control, 2 of the following precautions must be used: vasectomy, partner who uses hormonal contraception, tubal ligation, vaginal diaphragm, nonhormonal intrauterine device, condom, or sponge with spermicide.
* Females who are pregnant or lactating. A negative serum pregnancy test must be confirmed prior to the first dose of trial medication for all female subjects.
* Subjects presenting with a first episode of schizophrenia based on the clinical judgment of the investigator.
* Subjects who have received continuous medication therapy to treat schizophrenia for less than 6 months prior to the drug-free interval.
* Subjects with schizophrenia who are considered resistant/refractory to antipsychotic treatment by history, who have a history of failure to clozapine, or who are responsive only to clozapine treatment.
* Subjects with a current DSM-IV-TR Axis I diagnosis other than schizophrenia including MDD, bipolar disorder, delirium, dementia, amnestic, or other cognitive disorders or subjects with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder.
* Subjects who, in the opinion of the investigator, cannot be rated reliably on the battery of movement rating scales required by the protocol.
* Subjects with a significant risk of violent behavior, a significant risk of committing suicide based on history or investigator's judgment, or who have attempted suicide within 2 years of cohort assignment.
* Subjects with clinically significant tardive dyskinesia at enrollment.
* Subjects who experience clinical deterioration during the drug-free interval, such that they require prohibited rescue therapy, will not meet the trial criteria and will be replaced.
* Subjects who experienced an acute exacerbation requiring hospitalization within 3 months prior to the Screening Visit or between the Screening and Baseline Visits.
* Subjects who experienced an acute exacerbation requiring change in antipsychotic medication (with reference to drug or dose) within the last 4 weeks prior to baseline.
* Subjects who have a history of myocardial infarction, hypertension, or diabetes or who have evidence of other medical conditions that would expose them to an undue risk of a significant AE or interfere with assessments of safety or efficacy during the course of the trial, including, but not limited to, hepatic, renal, respiratory, cardiovascular, endocrine, neurologic, hematologic, or immunologic disease. The medical monitor must be contacted to discuss any such condition prior to cohort assignment.
* Subjects who have any of the following neurologic diagnoses, whether under treatment or not, whether stable or not: migraine, epilepsy, Parkinson's disease, Alzheimer's disease, multiple sclerosis, residual of stroke, transient cerebral ischemic attacks, cerebral palsy, or any condition that requires intermittent or maintenance treatment or which is manifested by any abnormality on neurologic examination. A subject with tardive dyskinesia or other nonclinically significant symptoms of EPS due solely to the current or prior use of antipsychotic medications is not excluded by this criterion. Single-nerve peripheral palsies are also not excluded by this criterion: eg, Bell's palsy or radial-nerve palsy or fixed residuals from traumatic injury.

History of or current hepatitis or acquired immunodeficiency syndrome or carriers of HBsAg and/or anti-HCV or HIV antibodies.

* Subjects with a history of thyroid pathology (unless the condition has been stabilized with medications for at least the past 3 months) and/or abnormal thyroid laboratory results.
* Subjects with a history of neuroleptic malignant syndrome.
* Subjects with a history of seizure disorder.
* Subjects who meet DSM-IV-TR criteria for substance dependence within 6 months prior to cohort assignment (excluding caffeine and nicotine), including alcohol and benzodiazepines, and/or a positive alcohol (breath or urine) test or a positive urine screen for drugs of abuse. (In the case where a subject had a positive screen for stimulants and/or marijuana and was therefore excluded, the medical monitor should be contacted to determine if rescreening is an option.)
* Subjects who had any major surgery, any blood transfusion, or donated blood or plasma within 30 days prior to enrollment.
* The following laboratory test, vital sign, and ECG results are exclusionary:

  1. Platelets <= 75,000/mm3
  2. Hemoglobin <= 9 g/dL
  3. Neutrophils, absolute <= 1000/mm3
  4. AST > 2 times upper limit of normal
  5. ALT > 2 times upper limit of normal
  6. Creatinine >= 2 mg/dL
* Subjects with electrolytes outside of the normal range will not be enrolled in the trial without prior review and approval from the medical monitor.
* Subjects who have sitting (performed first) or supine blood pressure, after resting for >= 3 minutes, higher than 140/90 mmHg or lower than 100/50 mmHg. Upon standing from the supine position, subjects who have a fall in systolic blood pressure >= 20 mmHg or a fall in diastolic blood pressure >= 10 mm Hg after 1 to 3 minutes in the standing position. (Any repeated out-of-range values not deemed clinically significant need to be discussed with the medical monitor to determine eligibility.)
* Subjects who have a supine pulse rate, after resting for >= 3 minutes, outside the range of 40 to 90 bpm.
* Subjects with any ECG abnormality at Screening, prior to dosing, will be excluded, including but not limited to, a PR interval > 220 msec, QRS interval > 110 msec, QTc > 450 msec, QTcF > 450 msec, QTcB > 450 msec or the increase in QTcB is considered significant by the investigator, abnormal U waves, or other minor ST-T wave changes which are considered clinically significant.
* Prohibited concomitant medications/therapies used for the following time period prior to Day -1 and for the duration of the trial include:
* Antipsychotics

  1. Use of oral antipsychotics within 21 days prior to Day -1;
  2. Use of long-acting injectable antipsychotics within 6 months.
* Anxiolytics and Sleep Aids

  1) Regular use of benzodiazepines for 2 weeks (lorazepam [<= 6 mg daily up to 48 hours prior to PK and PD assessments] can be used as rescue therapy during the 21 days prior to Day -1 and [<= 4 mg daily up to 48 hours prior to PK and PD assessments or up to 24 hours prior to the completion of the EPS rating scales or C-SSRS] during the treatment period).
* Mood Stabilizers

  1) Use of lamotrigine within 14 days.
* Selective Serotonin Reuptake Inhibitors

  1. Use of Prozac within 28 days;
  2. Use of Paxil within 14 days;
  3. Use of Zoloft, Luvox, or Celexa within 7 days.
* Serotonin and Norepinephrine Reuptake Inhibitors

  1. Use of Effexor within 3 days;
  2. Use of duloxetine within 14 days.
* Other

  1. Use of Symbyax within 28 days;
  2. Use of CYP2D6 or CYP3A4 inhibitors or CYP3A4 inducers within 14 days;
  3. Use of electroconvulsive therapy within 2 months.
* Use and discontinuation of any other therapy (prescription medication, over-the counter, herbal medication, or vitamins) not listed above must be approved by the sponsor and the medical monitor.
* Subjects who received brexpiprazole in a prior clinical trial.
* Subjects who received any investigational agent in a clinical trial within 90 days prior to Screening.
* Consumption of alcohol and/or food and beverages containing methylxanthines, grapefruit, grapefruit juice, Seville oranges, or Seville orange juice within 72 hours prior to dosing and for the duration of the trial.
* Subjects who are heavy smokers (ie, > 21 cigarettes per day). Other
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious disease) illness must not be enrolled into this trial.
* Subjects with a history of allergy to more than one class of medications.
* Any subject who, in the opinion of the investigator, should not participate in the trial.
* A history of difficulty in donating blood.
* Exposure to any substances known to stimulate hepatic microsomal enzymes within 30 days prior to Screening through the end of the trial (eg, occupational exposure to pesticides, organic solvents).
* Additionally, subjects who meet the following imaging exclusion criteria will not be included in this trial:

  1. Subjects who suffer from claustrophobia.
  2. Subjects with MRI-incompatible implants and other contraindications for MRI, such as pacemaker, artificial joints, nonremovable body piercings, tattoos larger than 1 cm in diameter, metal fragments, claustrophobia, etc.
  3. Subjects who have received a diagnostic or therapeutic radiopharmaceutical within 7 days prior to participation in this trial.
  4. Participation in other research trials involving ionizing radiation within 1 year of the PET scans that would cause the subject to exceed the yearly dose limits for normal subjects.
  5. Subjects with history of IV drug use which would prevent venous access for PET tracer injection.
  6. Severe motor problems that prevent the subject from lying still for PET and MRI.
  7. Subjects who complain of chronic pain (eg, as the result of rheumatoid arthritis).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2013-09; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Derived] Girgis RR, Forbes A, Abi-Dargham A, Slifstein M. A positron emission tomography occupancy study of brexpiprazole at dopamine D2 and D3 and serotonin 5-HT1A and 5-HT2A receptors, and serotonin reuptake transporters in subjects with schizophrenia. Neuropsychopharmacology. 2020 Apr;45(5):786-792. doi: 10.1038/s41386-019-0590-6. Epub 2019 Dec 17. PMID 31847007

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Phase 1, single center, open-label trial of up to 12 enrolled participants.
Pre-assignment Details: Participants were at the inpatient unit in the New York State Psychiatric Institute between Days -22 and -2. Participants remained inpatient during the drug-free interval at the principal investigator's discretion.
Groups:
- Cohort 1 - Brexpiprazole 4 mg: Participants in cohort 1 received 1 milligram (mg) tablet of brexpiprazole once daily on Days 1 to 3 and 4-mg tablet of brexpiprazole once daily on Days 4 to 10.
- Cohort 2 - Brexpiprazole 1 mg: Participants in cohort 2 received 1-mg tablet of brexpiprazole once daily on Days 1 to 10.
- Cohort 3 - Brexpiprazole 4 mg: Participants in cohort 3 received 1- to 4-mg dose of brexpiprazole (at the study physician's discretion) once daily on Days 1 to 3 and 4-mg tablet of brexpiprazole once daily on Days 4 to 10.
Period: Overall Study
Arm/Group | Cohort 1 - Brexpiprazole 4 mg | Cohort 2 - Brexpiprazole 1 mg | Cohort 3 - Brexpiprazole 4 mg
Started | 4 | 4 | 4
Completed | 4 | 4 | 3
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 - Brexpiprazole 4 mg: Participants in cohort 1 received 1-mg tablet of brexpiprazole once daily on Days 1 to 3 and 4-mg tablet of brexpiprazole once daily on Days 4 to 10.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Brexpiprazole 4 mg | Cohort 2 - Brexpiprazole 1 mg | Cohort 3 - Brexpiprazole 4 mg | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.3 (4.4) | 40.8 (11.9) | 45 (6.9) | 41.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 5
  Male | 1 | 3 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage Dopamine D2/D3 Receptor Occupancy
Description: Dopamine receptor occupancy measured using the radiotracer [11C]-(+)-PHNO in low and high dose. The binding of brexpiprazole to the D2/D3 receptors were assessed by comparing the binding potential from the Baseline scan (prior to treatment) to that of Day 10 (after treatment). The D2/D3 receptors following administration of a 1- and 4-mg doses of brexpiprazole were assessed and the occupancy estimates were averaged across brain regions 4 hours post-last dose on Day 10.
Time Frame: Baseline to 4 hours post-last dose on Day 10
Population: The positron emission tomography (PET) analysis included all participants who had both the Baseline and Day 10 PET scans performed.
Measure: Mean (Standard Deviation); unit: percentage occupancy
Groups:
- Brexpiprazole 1mg: Participants received 1-mg tablet of brexpiprazole once daily on Days 1 to 10.
- Brexpiprazole 4 mg: Participants received 1-mg brexpiprazole once daily on Days 1 to 3 and 4-mg tablet of brexpiprazole once daily on Days 4 to 10.
Arm/Group | Brexpiprazole 1mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 4 | 4
percentage occupancy
  6-region model (D2 receptor) | 36 (16) | 59 (5)
  6-region model (D3 receptor) | 2 (3) | 13 (10)
  8-region model (D2 receptor) | 27 (25) | 67 (15)
  8-region model (D3 receptor) | 1 (2) | 31 (8)

2. Primary Outcome: Change in Percentage 5-HT1A Receptor Occupancy
Description: Mean (±SD) Serotonin 5-HT1A Receptor Occupancy Using the Radiotracer [11C]CUMI101 in high dose only. In cohorts 1, 2 and 3, the binding of brexpiprazole to the 5-HT1A receptors was assessed by comparing the binding potential from the Baseline scan (prior to treatment) to that of Day 10 (after treatment). The 5-HT1A receptors following administration of a 4-mg dose of brexpiprazole was assessed and the occupancy estimates were averaged across brain regions 4 hours post-last dose on Day 10.
Time Frame: Baseline to 4 hours post-last dose on Day 10
Population: The PET analysis included all participants who had both the Baseline and Day 10 PET scans performed.
Measure: Mean (Standard Deviation); unit: percentage occupancy
Groups:
- Brexpiprazole 4mg: Participants received 1- to 4-mg dose of brexpiprazole (at the study physician's discretion) once daily on Days 1 to 3 and 4-mg tablet of brexpiprazole once daily on Days 4 to 10.
Arm/Group | Brexpiprazole 4mg
Number analyzed (Participants) | 4
percentage occupancy | 4 (6)

3. Primary Outcome: Change in Percentage 5-HT2A Receptor Occupancy
Description: Mean (±SD) Serotonin 5-HT2A Receptor Occupancy Using the Radiotracer [11C]MDL100907 (in low and high dose). The 5-HT2A receptors following administration of 1- and 4-mg doses of brexpiprazole were assessed and the occupancy estimates were averaged across brain regions 4 hours post-last dose on Day 10.
Time Frame: Baseline and 4 hours post-last dose on Day 10
Population: The PET analysis included all participants who had both the Baseline and Day 10 PET scans performed.
Measure: Mean (Standard Deviation); unit: percentage occupancy
Arm/Group | Brexpiprazole 1mg | Brexpiprazole 4 mg
Number analyzed (Participants) | 4 | 4
percentage occupancy | 28 (10) | 45 (7)

4. Primary Outcome: Change in Occupancy at Serotonin Transporter (SERT)
Description: Mean (±SD) SERT Occupancy Using the Radiotracer [11C]DASB in high dose only. Occupancy estimates were averaged across brain regions 4 hours post-last dose.
Time Frame: Baseline to 4 hours post-last dose on Day 10
Population: The PET analysis included all participants who had both the Baseline and Day 10 PET scans performed.
Measure: Mean (Standard Deviation); unit: percentage occupancy
Groups:
- Brexpiprazole 4mg: Participants in cohort 3 received 1- to 4-mg dose of brexpiprazole (at the study physician's discretion) once daily on Days 1 to 3 and 4-mg tablet of brexpiprazole once daily on Days 4 to 10.
Arm/Group | Brexpiprazole 4mg
Number analyzed (Participants) | 4
percentage occupancy | -3 (15)

5. Secondary Outcome: Area Under the Concentration-time Curve (AUCτ) During a Dosing Interval at Steady-state for Brexpiprazole and Its Metabolite DM-3411
Description: AUC during a dosing interval at steady-state for brexpiprazole and its metabolite DM-3411. Days 1 and 9: predose (within 15 minutes prior to dosing) Day 10: predose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 8, and 12 hours post-last dose.
Time Frame: Baseline to Day 10
Population: The PK analysis included participants who had valid measurements (per clinical pharmacology). Blood samples were collected on Days 1 and 9 at predose and Day 10 at predose and at 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-last dose or at early termination (ET).
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Cohort 1 - Brexpiprazole 4mg: Participants in Cohort 1 received 1-mg tablet of brexpiprazole once daily on Days 1 to 3 and 4-mg tablet of brexpiprazole once daily on Days 4 to 10.
- Cohort 2 - Brexpiprazole 1mg: Participants in Cohort 2 received one 1-mg tablet of brexpiprazole once daily on Days 1 to 10.
- Cohort 3 - Brexpiprazole 4 mg: Participants in Cohort 3 received one 1- to 4-mg dose of brexpiprazole (at the investigator's discretion) once daily on Days 1 to 3 and one 4-mg tablet of brexpiprazole once daily on Days 4 to 10.
Arm/Group | Cohort 1 - Brexpiprazole 4mg | Cohort 2 - Brexpiprazole 1mg | Cohort 3 - Brexpiprazole 4 mg
Number analyzed (Participants) | 4 | 4 | 4
hr*ng/mL
  Brexpiprazole | 2520 (1290) | 716 (118) | 1410 (352)
  DM-3411 | 807 (205) | 329 (227) | 761 (397)

6. Secondary Outcome: Peak (Maximal) Concentration of Drug in Plasma (Cmax) for Brexpiprazole and Its Metabolite DM-3411
Description: (Cmax) Days 1 and 9: predose (within 15 minutes prior to dosing) Day 10: predose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 8, and 12 hours post-last dose.
Time Frame: Baseline to Day 10
Population: The PK analysis included participants who had valid measurements (per clinical pharmacology). Blood samples were collected on Days 1 and 9 at predose and Day 10 at predose and at 1, 2, 3, 4, 5, 6, 8, 12, and 24 hours post-last dose or at ET.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cohort 1 - Brexpiprazole 4mg: Participants in cohort 1 received 1-mg of brexpiprazole once daily on Days 1 to 3 and 4-mg tablet of brexpiprazole once daily on Days 4 to 10.
- Cohort 2- Brexpiprazole 1mg: Participants in cohort 2 received 1-mg tablet of brexpiprazole once daily on Days 1 to 10.
- Cohort 3 - Brexpiprazole 4mg: Participants in cohort 3 received 1- to 4-mg dose of brexpiprazole (at the study physician's discretion) once daily on Days 1 to 3 and 4-mg tablet of brexpiprazole once daily on Days 4 to 10.
Arm/Group | Cohort 1 - Brexpiprazole 4mg | Cohort 2- Brexpiprazole 1mg | Cohort 3 - Brexpiprazole 4mg
Number analyzed (Participants) | 4 | 4 | 3
ng/mL
  Brexpiprazole | 126 (58.3) | 46.5 (7.47) | 70.9 (18.8)
  DM-3411 | 37.1 (10.8) | 17.3 (10.4) | 35.7 (18.6)

7. Secondary Outcome: Apparent Clearance of Drug From Plasma After Extravascular Administration (CL/F; Only Brexpiprazole)
Description: PK parameter - CL/F was assessed for brexpiprazole only. Days 1 and 9: predose (within 15 minutes prior to dosing) Day 10: predose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 8, and 12 hours post-last dose.
Time Frame: Baseline to Day 10
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mL/hr
Groups:
- Cohort 1 - Brexpiprazole 4 mg: Participants in cohort 1 received 1-mg of brexpiprazole once daily on Days 1 to 3 and 4-mg tablet of brexpiprazole once daily on Days 4 to 10.
Arm/Group | Cohort 1 - Brexpiprazole 4 mg | Cohort 2 - Brexpiprazole 1mg | Cohort 3 - Brexpiprazole 4mg
Number analyzed (Participants) | 4 | 4 | 4
mL/hr | 1960 (960) | 1420 (242) | 2970 (831)

8. Secondary Outcome: Time to Maximum (Peak) Plasma Concentration (Tmax) for Brexpiprazole and Its Metabolite DM-3411
Description: Tmax for brexpiprazole and its metabolite DM-3411. Days 1 and 9: predose (within 15 minutes prior to dosing) Day 10: predose (within 15 minutes prior to dosing) and 1, 2, 3, 4, 5, 6, 8, and 12 hours post-last dose.
Time Frame: Baseline to Day 10
Population: as for outcome 6
Measure: Median (Full Range); unit: hour
Groups:
- Cohort 3 - Brexpiprazole 4mg: Participants in cohort 3 received once 1- to 4-mg dose of brexpiprazole (at the study physician's discretion) once daily on Days 1 to 3 and one 4-mg tablet of brexpiprazole once daily on Days 4 to 10.
Arm/Group | Cohort 1 - Brexpiprazole 4mg | Cohort 2 - Brexpiprazole 1mg | Cohort 3 - Brexpiprazole 4mg
Number analyzed (Participants) | 4 | 4 | 4
hour
  Brexpiprazole | 1.92 [0.00 to 2.92] | 1.50 [0.93 to 1.93] | 4.87 [3.10 to 6.00]
  DM-3411 | 2.42 [0.00 to 24.08] | 1.51 [0.00 to 11.92] | 11.87 [3.10 to 24.00]

9. Secondary Outcome: Mean Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Score
Description: The AIMS Scale was an extrapyramidal symptoms (EPS) rating scale. The AIMS is a 12 item scale. The first 10 items e.g. facial and oral movements (items 1-4), extremity movements (items 5 and 6), trunk movements (item 7), investigators global assessment of dyskinesia (items 8 to 10). The first 10 items are rated from 0 to 4 (0=best, 4=worst). Items 11 and 12, related to dental status, have dichotomous responses, 0=no and 1=yes. The AIMS Total Score is the sum of the ratings for the first seven items. The possible total scores are from 0 to 28, with a higher score indicating worse outcome. Last Visit is the last scheduled post-baseline evaluation including early termination evaluation.
Time Frame: Baseline to Day 6, 11 and Last Visit
Population: The safety population included all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Cohort 2 - Brexpiprazole 1mg: Participants in cohort 2 received 1-mg tablet of brexpiprazole once daily on Days 1 to 10.
- Cohort 3 Brexpiprazole 4mg: Participants in cohort 3 received 1- to 4-mg dose of brexpiprazole (at the study physician's discretion) once daily on Days 1 to 3 and 4-mg tablet of brexpiprazole once daily on Days 4 to 10.
Arm/Group | Cohort 1 - Brexpiprazole 4mg | Cohort 2 - Brexpiprazole 1mg | Cohort 3 Brexpiprazole 4mg
Number analyzed (Participants) | 4 | 4 | 4
Units on a scale
  Day 6 | 0 (0) | 0 (0) | 0.3 (0.5)
  Day 11 | 0 (0) | 0 (0) | 0 (0)
  Last Visit | 0 (0) | 0 (0) | 0 (0)

10. Secondary Outcome: Mean Change From Baseline in Simpson-Angus Scale (SAS) Total Score
Description: The SAS is a rating scale used to measure EPS. The SAS scale consists of a list of 10 symptoms of parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia), with each item rated from 0 to 4, with 0 being normal and 4 being the worst. The SAS Total score is sum of ratings for all 10 items, with possible Total scores from 0 to 40, with higher scores indicating worse outcome. Last Visit is the last scheduled post-baseline evaluation including early termination evaluation.
Time Frame: Baseline to Day 6, 11 and Last Visit
Population: The safety population included all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on scale
Groups:
- Cohort 2- Brexpiprazole 1mg: Participants in cohort 2 received one 1-mg tablet of brexpiprazole once daily on Days 1 to 10.
- Cohort 3 Brexpiprazole 4mg: Participants in cohort 3 received once 1- to 4-mg dose of brexpiprazole (at the study physician's discretion) once daily on Days 1 to 3 and one 4-mg tablet of brexpiprazole once daily on Days 4 to 10.
Arm/Group | Cohort 1 - Brexpiprazole 4mg | Cohort 2- Brexpiprazole 1mg | Cohort 3 Brexpiprazole 4mg
Number analyzed (Participants) | 4 | 4 | 4
Units on scale
  Day 6 | 0.3 (0.5) | 0 (0) | -0.3 (1.3)
  Day 11 | 0 (0) | 0 (0) | -0.7 (1.2)
  Last Visit | 0 (0) | 0 (0) | -0.5 (1.0)

11. Secondary Outcome: Mean Change From Baseline in Barnes Akathisia Rating Scale (BARS) Score
Description: The BARS consisted of 4 items related to akathisia: objective observation of akathisia by the study physician, subjective feelings of restlessness by the participant, participant distress due to akathisia, and global evaluation of akathisia. The first 3 items were rated on a 4-point scale, with a score of 0 = absence of symptoms and a score of 3 = severe condition. The global clinical evaluation were made on a 6-point scale, (0=absent, 1=questionable, 2=mild, 3=moderate, 4=marked, 5=severe). To complete this scale, participants were observed while they were seated and then stood for a minimum of 2 minutes in each position. Symptoms observed in other situations (e.g., while engaged in neutral conversation or engaged in activity on the ward) may also be rated. Subjective phenomena were to be elicited by direct questioning. The BARS total score (when combined) ranged from 0 to 18, with higher values indicating a severe condition.
Time Frame: Baseline to Day 6, 11 and Last Visit
Population: The safety population included all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort 1 - Brexpiprazole 4mg | Cohort 2- Brexpiprazole 1mg | Cohort 3 Brexpiprazole 4mg
Number analyzed (Participants) | 4 | 4 | 4
Units on a scale
  Day 6 | 0.5 (1.0) | 0 (0) | 0.5 (1.0)
  Day 11 | 0.5 (1.0) | 0 (0) | 0.0 (0.0)
  Last Visit | 0.5 (1.0) | 0 (0) | 0.0 (0.0)

12. Secondary Outcome: Percentage of Participants Who Reported at Least One Occurrence of Suicidality, Suicidal Behavior and Suicidal Ideation on the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. Suicidality was defined as reporting at least one occurrence of any suicidal behavior or suicidal ideation. Suicidal behavior was defined as reporting any type of suicidal behaviors (actual attempt, interrupted attempt, aborted attempt, and preparatory acts or behavior). The suicidal ideation intensity total score is the sum of intensity scores of 5 items (frequency, duration, controllability, deterrents, and reasons for ideation). The score of each intensity item ranges from 0 (none) to 5 (worst) which leads to the range of the total score from 0 to 25, with a higher score indicating a worse outcome. A missing score of any item resulted in a missing total score. If no suicidal ideation was reported, a score of 0 was given to the intensity scale. Last Visit is last scheduled post-baseline evaluation including early termination evaluation.
Time Frame: Baseline to Last Visit
Population: The safety population included all participants who received at least one dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 - Brexpiprazole 4mg | Cohort 2- Brexpiprazole 1mg | Cohort 3 Brexpiprazole 4mg
Number analyzed (Participants) | 4 | 4 | 4
Percentage of participants
  Suicidality | 0 | 0 | 0
  Suicidal behaviour | 0 | 0 | 0
  Suicidal Ideation | 0 | 0 | 0

13. Secondary Outcome: Mean Change From Baseline in Positive and Negative Symptom Scale (PANSS) Total Score
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS total score was the sum of the rating scores for 7 positive scale items, 7 negative scale items, and 16 general psychopathology scale items from the PANSS panel. The PANSS total score ranged from 30 (best possible outcome) to 210 (worst possible outcome). Last Visit is the last scheduled post-baseline evaluation including early termination evaluation.
Time Frame: Baseline to Day 6, 11 and Last Visit
Population: The safety sample included participants that are administered at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort 1 - Brexpiprazole 4mg | Cohort 2 - Brexpiprazole 1mg | Cohort 3 - Brexpiprazole 4mg
Number analyzed (Participants) | 4 | 4 | 4
Units on a scale
  Day 6 | -4.0 (7.4) | 0.3 (4.0) | -2.0 (3.9)
  Day 11 | -1.5 (5.2) | 6.0 (11.1) | -4.0 (10.5)
  Last Visit | -1.5 (5.2) | 6.0 (11.1) | -3.0 (8.7)

14. Secondary Outcome: Mean Change From Baseline in PANNS Positive Subscale Score
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS positive subscale score was the sum of the rating scores for the 7 positive scale items from the PANSS panel. The 7 positive symptom constructs are delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. The PANSS Positive Subscale ranges from 7 (absence of symptoms) to 49 (extremely severe symptoms). Last Visit is the last scheduled post-baseline evaluation including early termination evaluation.
Time Frame: Baseline to Day 6, 11 and Last Visit
Population: The safety population included all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort 1 - Brexpiprazole 4mg | Cohort 2- Brexpiprazole 1mg | Cohort 3 Brexpiprazole 4mg
Number analyzed (Participants) | 4 | 4 | 4
Units on a scale
  Day 6 | -0.8 (1.0) | 0.0 (2.0) | -0.8 (3.9)
  Day 11 | 0.5 (1.0) | 0.5 (6.1) | -2.7 (7.5)
  Last Visit | 0.5 (1.0) | 0.5 (6.1) | -2.0 (6.3)

15. Secondary Outcome: Mean Change From Baseline in PANSS Negative Subscale Score
Description: The PANSS consisted of three subscales: a total of 30 symptom constructs. For each symptom construct, severity was rated on a 7-point scale, with a score of 1 (absence of symptoms) and a score of 7 (extremely severe symptoms). The PANSS negative subscale score was the sum of the rating scores for the 7 negative scale items from the PANSS panel. The 7 negative symptom constructs: blunted affect, emotional withdrawal, poor rapport, passive apathetic withdrawal, difficulty in abstract thinking, lack of spontaneity and flow of conversation, stereotyped thinking. The PANSS Negative Subscale ranges from 7 (absence of symptoms) to 49 (extremely severe symptoms). Last Visit is the last scheduled post-baseline evaluation including early termination evaluation.
Time Frame: Baseline to Day 6, 11 and Last Visit
Population: The safety population included all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort 1 - Brexpiprazole 4mg | Cohort 2- Brexpiprazole 1mg | Cohort 3 Brexpiprazole 4mg
Number analyzed (Participants) | 4 | 4 | 4
Units on a scale
  Day 6 | -2.5 (4.4) | 1.0 (1.0) | 0.3 (1.0)
  Day 11 | -1.5 (2.4) | 0.5 (3.0) | -0.3 (3.2)
  Last Visit | -1.5 (2.4) | 0.5 (3.0) | -0.3 (2.6)

16. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score
Description: The severity of illness for each participant was rated using the CGI-S scale. To assess CGI-S, the study physician answered the following question: "Considering your total clinical experience with this particular population, how mentally ill is the participant at this time?" Response choices included: 0 = not assessed; 1 = normal, not ill at all; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill participants. Last Visit is the last scheduled post-baseline evaluation including early termination evaluation.
Time Frame: Baseline to Day 6, 11 and Last Visit
Population: The safety population included all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort 1 - Brexpiprazole 4mg | Cohort 2- Brexpiprazole 1mg | Cohort 3 Brexpiprazole 4mg
Number analyzed (Participants) | 4 | 4 | 4
Units on a scale
  Day 6 | 0.3 (0.5) | 0.0 (0.0) | 0.8 (1.0)
  Day 11 | 0.5 (1.0) | 0.0 (0.0) | 1.0 (1.0)
  Last Visit | 0.5 (1.0) | 0.0 (0.0) | 0.8 (1.0)

17. Secondary Outcome: Mean Change From Baseline in Clinical Global Impression-Improvement (CGI-I) Score
Description: The efficacy of trial medication were rated for each participant using the CGI-I scale. The study physician must rate the participant's total improvement whether or not it is due entirely to drug treatment. All responses were compared to the participant's condition at baseline. Response choices include: 0 = not assessed; 1 =very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 =minimally worse; 6 = much worse; and 7 = very much worse. Last Visit is the last scheduled post-baseline evaluation including early termination evaluation.
Time Frame: Baseline to Day 6, 11 and Last Visit
Population: The safety population included all participants who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cohort 1 - Brexpiprazole 4mg | Cohort 2- Brexpiprazole 1mg | Cohort 3 Brexpiprazole 4mg
Number analyzed (Participants) | 4 | 4 | 4
Units on a scale
  Day 6 | 4.0 (0.0) | 4.0 (0.0) | 4.0 (0.0)
  Day 11 | 3.5 (1.0) | 3.8 (0.5) | 2.7 (1.2)

ADVERSE EVENTS:
Time Frame: Adverse events were reported once the informed consent was signed, throughout the 10-day treatment period until the safety follow-up via telephone 30 (+2) days post-last dose of study medication.
Groups:
- Cohort 1 - Brexpiprazole 4 mg: Participants in cohort 1 received one 1-mg of brexpiprazole once daily on Days 1 to 3 and one 4-mg tablet of brexpiprazole once daily on Days 4 to 10.
- Cohort 2 - Brexpiprazole 1 mg: Participants in cohort 2 received one 1-mg tablet of brexpiprazole once daily on Days 1 to 10.
- Cohort 3 - Brexpiprazole 4 mg: Participants in cohort 3 received once 1- to 4-mg dose of brexpiprazole (at the study physician's discretion) once daily on Days 1 to 3 and one 4-mg tablet of brexpiprazole once daily on Days 4 to 10.
Arm/Group | Cohort 1 - Brexpiprazole 4 mg | Cohort 2 - Brexpiprazole 1 mg | Cohort 3 - Brexpiprazole 4 mg
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 2/4 | 3/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Brexpiprazole 4 mg (N=4) | Cohort 2 - Brexpiprazole 1 mg (N=4) | Cohort 3 - Brexpiprazole 4 mg (N=4)
Blepharospasm (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Dental carries (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Akathisia (Nervous system disorders) | 1 | 0 | 1
Sedation (Nervous system disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less